CLINICAL TRIAL: NCT05728489
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous and Subcutaneous Multiple Rising Doses of BI 765250 Versus Placebo in Trial Participants With Moderate to Severe Plaque Psoriasis (Double-blind, Randomised, Placebo-controlled, Parallel-group Design)
Brief Title: A Study to Test How Well Different Doses of BI 765250 Are Tolerated by People With a Skin Disease Called Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1474-0002; 2021-006280-25 (EudraCT Number); 2024-512420-10-00 (Other: CTIS); U1111-1308-0095 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BI 765250 very low dose group (Experimental)
  Interventions: Drug: BI 765250
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 765250 low dose group (Experimental)
  Interventions: Drug: BI 765250
- BI 765250 medium dose group (Experimental)
  Interventions: Drug: BI 765250
- BI 765250 high dose group (Experimental)
  Interventions: Drug: BI 765250
- BI 765250 very high dose group (Experimental)
  Interventions: Drug: BI 765250

INTERVENTIONS:
Drug: BI 765250 — BI 765250
  Arms: BI 765250 high dose group; BI 765250 low dose group; BI 765250 medium dose group; BI 765250 very high dose group; BI 765250 very low dose group
Drug: Placebo — placebo
  Arms: Placebo group

SUMMARY:
This study is open to adults with plaque psoriasis. The main purpose of this study is to find out whether people with plaque psoriasis can tolerate a medicine called BI 765250. Another purpose is to check whether BI 765250 can improve participants' skin condition.

Participants are divided into 5 groups. Each group gets a different dose of BI 765250 or placebo as an infusion or injection for 12 weeks. Placebo infusions and injections look like BI 765250 but do not contain any medicine. It is decided by chance, who gets BI 765250 and who gets placebo. During the first 2 weeks, participants get the study medicine as an infusion into a vein once a week. Afterwards, they get the study medicine as an injection under the skin every 2 or 4 weeks. In total, every participant gets up to 5 injections.

Participants are in the study for about 8 months. During this time, they visit the study site 23 times. On 2 of the visits, participants stay overnight at the study site, once for 2 nights and once for 1 night. The doctors collect information on any health problems of the participants. They also regularly check participants' skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential and male participants
* Age 18 to 75 years (both inclusive) at the time of informed consent
* Diagnosis of chronic plaque psoriasis for at least 6 months prior to randomisation, as confirmed by their medical record or history
* Moderate to severe plaque psoriasis, as defined by:

  * Body surface area (BSA) ≥5% and <30%
  * Static Physician's Global Assessment (sPGA) ≥3
  * Target lesions suitable for skin biopsy
* Body mass index (BMI) <35 kg/m2
* Male participants able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the participant information
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Non-plaque forms of psoriasis, current drug-induced psoriasis, or active ongoing inflammatory diseases other than psoriasis that might confound trial evaluations
* Major surgery (major according to the investigator's assessment, e.g. hip replacement) performed within 16 weeks prior to randomisation or planned during the trial (i.e. until the End of Study Visit)
* Women of childbearing potential (WOCBP), breastfeeding women, and men unwilling or unable to use highly effective methods of birth control
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening
* Live or attenuated vaccination ≤6 weeks prior to randomisation, or any plan to receive a live vaccination during the conduct of this trial until the End of Treatment Visit
* Participants who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Hepatic/renal impairment:

  * Hepatic impairment defined as >3-fold Upper Limit of Normal (ULN) elevation in AST or ALT or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin. Trial participants with Gilbert´s syndrome can be included unless total bilirubin elevation was >5-fold ULN at screening visit and unless proportions of bilirubin fractions are inconsistent with diagnosis of Gilbert´s syndrome.
  * Renal impairment defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
* Currently enrolled in an investigational drug or device study, or use of any investigational drug or device within 4 weeks prior to randomisation or 5 half-lives of the drug (whichever is longer) Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of any adverse events | Up to Day 239

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in serum at steady state over a uniform dosing interval τ (Cmax,ss) | Up to Day 85
Time from last dosing to maximum concentration of the analyte in serum at steady state (tmax,ss) | Up to Day 85
Area under the concentration-time curve of the analyte in serum at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to Day 85
Absolute change from baseline in the Static Physician's Global Assessment (sPGA) x Body Surface Area (BSA) score | At baseline and at week 12
Percentage change from baseline in the sPGA x BSA score | At baseline and at week 12

CONTACTS AND LOCATIONS:
Locations (5):
- MBAL Sveta Sofia, Sofia, Bulgaria
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- Clinical Republican Hospital "Timofei Mosneaga", Chisinau, Moldova
- Romania (2):
  - MONZA Medical Center, Bucharest
  - Emergency County Hospital, Arensia EM, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com